CLINICAL TRIAL: NCT05372757
Title: Partial Heart Transplantation for Severe Pediatric Semilunar Valve Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00114653
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Semilunar Heart Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Partial Heart Transplantation Arm (Experimental)
  Interventions: Procedure: Partial Heart Transplantation

INTERVENTIONS:
Procedure: Partial Heart Transplantation — The donor heart will be recovered and the new heart valve will be removed from this heart by the clinical team. The child will be scheduled for an emergent operation once the donor heart valve is deemed acceptable. The child will have general anesthesia during surgery. This is a state of unconsciousness, which is carefully controlled by the anesthesiologist with a mixture of very potent drugs, to prevent or lessen pain. The child will have a partial heart transplant using the donated heart valve to replace the dysfunctional heart valve. Expected hospital stay will range from weeks to months. The medical care after surgery is performed by the child's clinical team. This type of re-operation could similarly be required after a standard heart valve replacement.

SUMMARY:
The long-term goal of this research initiative is to develop a new valve replacement option for neonates, infants and young children. The central hypothesis is that transplantation of a freshly isolated heart valve will be associated with superior outcomes compared to currently available options, including preserved cadaver valves, bioprosthetic tissue valves, or mechanical valves. This new operation has been named "partial heart transplantation".

The proposed study is a single-center, nonrandomized single arm pilot trial of "partial heart transplantation" in neonates, infants and young children who require semilunar heart valve replacement. This "first in man" trial seeks to determine whether valve replacement using partial heart transplant is feasible and safe. Primary aims are survival one year and five years following the procedure. The hypothesis is that, when compared to historical controls who have undergone homograft valve replacement, those undergoing partial heart transplantation will have equal or superior survival one year and five years following the procedure. Secondary aims are to assess growth and function of the transplanted valve. The hypothesis is that when compared to historical controls who have undergone conventional valve replacement, those undergoing partial heart transplantation will have valve growth that corresponds with somatic growth and superior valve function 1 year following the procedure. Up to five patients will be enrolled in this trial over three years.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 2 years of age who are referred for a cardiac operation that involves a primary semilunar valve replacement or children less than 2 years of age who are referred for a cardiac operation involves an initial replacement of a previously placed prior homograft, bioprosthetic, or mechanical valve in the aortic or pulmonary position.
* Deemed acceptable for partial heart transplantation based on the standard evaluation process used for orthotopic heart transplantation (see Appendix 1) Insurance approval.
* Written informed consent of both parents/guardians; if there is only one parent/guardian, consent from that individual will be adequate.

Exclusion Criteria:

* Absolute contraindications for orthotopic heart transplantation.
* Severe bilateral long segment pulmonary arterial hypoplasia
* Bilateral pulmonary vein stenosis
* <34 weeks corrected gestational age
* Persistent acidosis with a pH < 7.1
* Diagnosis of immune deficiency.
* Inability for the parent to understand English or Spanish.
* Failure to pass the following psychosocial evaluation:
* The candidate should reside within 4 hours traveling time from Medical University of South Carolina for a minimum of four to six months post-transplantation to assure careful follow-up
* The candidate's family should be capable of long-term supportive care of the child and be able to support the medical needs of the child in follow-up
* Parental (custodial) alcohol and/or substance abuse
* Documented parental (custodial) child abuse or neglect
* Parent (custodian) with cognitive/psychiatric impairment severe enough to limit comprehension of medical regimen
* Infectious Disease Exclusion Criteria
* Evidence of sepsis
* Hepatitis B surface antigenemia
* HIV positivity

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
The ability to perform the new operation in at least 1 patient per year for 3 years (averaged) after enrollment opens. | Duration of the study (3 years after enrollment opens).
  This is how feasibility will be measured. This will be answered as "yes" or "no".
Number of participants who achieve survival. | 6 months after all 5 subjects have been enrolled.
  Safety will primarily be defined as patient survival or re-operation or transcatheter reintervention on the transplanted valve at 6-month intervals, starting 6 months after the first subject undergoes a valve transplant, and continuing until 1 year after all 5 subjected have been enrolled.
Number of participants who achieve survival. | 1 year after all 5 subjects have been enrolled.
  Safety will primarily be defined as patient survival or re-operation or transcatheter reintervention on the transplanted valve at 6-month intervals, starting 6 months after the first subject undergoes a valve transplant, and continuing until 1 year after all 5 subjected have been enrolled.

SECONDARY OUTCOMES:
Valve annulus growth. | Every 6 months following the operation until child is old enough (18+ years) for mechanical prosthesis or date of death, whichever comes first.
  The valve annulus diameter will be measured using echocardiography in 2 planes at baseline (i.e., during postoperative hospitalization 5-10 days after surgery) and every 6 months following the operation. It is expected that the valve annulus diameter Z score will be relatively unchanged over time, which would reflect an absolute increase in valve annulus growth corresponding with an increase in body surface area.
The level of valve stenosis. | Every 6 months following the operation until child is old enough (18+ years) for mechanical prosthesis or date of death, whichever comes first.
  Mean valve stenosis will be assessed by transthoracic echocardiogram using pulse Doppler every 6 months following the operation.
The level of valve regurgitation. | Every 6 months following the operation until child is old enough (18+ years) for mechanical prosthesis or date of death, whichever comes first.
  Mean valve regurgitation will be assessed with color Doppler echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Taufiek Rajab, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rajab TK, Ochoa B, Zilinskas K, Kwon J, Taylor CL, Henderson HT, Savage AJ, Kavarana M, Turek JW, Costello JM. Partial heart transplantation for pediatric heart valve dysfunction: A clinical trial protocol. PLoS One. 2023 Feb 7;18(2):e0280163. doi: 10.1371/journal.pone.0280163. eCollection 2023. PMID 36749770